CLINICAL TRIAL: NCT00223600
Title: Special Turku Atherosclerosis Risk Factor Intervention Project for Children (STRIP)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Turku (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STRIP19902010; Academy of Finland (grant)
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2006-09-19 (Estimated); Status verified 2005-08

CONDITIONS: Atherosclerosis
Keywords: lipids; lipoproproteins; growth; neurological development; vascular wall; blood pressure; nutrient intake
MeSH Terms: conditions — Atherosclerosis

INTERVENTIONS:
Behavioral: Nutritional and life style counseling

SUMMARY:
1062 children at the age of 7 months and their families were randomized 1:1 in an intervention arm and a control arm. The intervention families has received child-oriented and individualized nutritional and life-style counseling that aims at decreasing child's exposure to the known environmental atherosclerosis risk factors. The controls children receive information as given at the well-baby clinics and in school health care of children and adolescents. The hypothesis is that the intervention children have healthier food habits and serum serum lipid and lipoprotein concentrations than the controls, fewer of them start smoking, and their physical activity level is higher than that of the controls.

DETAILED DESCRIPTION:
1062 children at the age of 7 months and their families were randomized 1:1 in an intervention arm and a control arm. The intervention families has received child-oriented and individualized nutritional and life-style counseling that aims at decreasing child's exposure to the known environmental atherosclerosis risk factors. The controls children receive information as given at the well-baby clinics and in school health care of children and adolescents. The hypothesis is that the intervention children have healthier food habits and serum serum lipid and lipoprotein concentrations than the controls, fewer of them start smoking, and their physical activity level is higher than that of the controls. We further hypothesised that the life-style intervention had no adverse mental or somatic effects on the children. Intima-media thickness of the carotid and brachial arterias and aorta and vasodilatation of the brachial artery induced by endogenous NO production have been also been measures at 2-year intervals since the age of 11 years. Recruitment to the study began in 1990 and continued for 2 years. The children are now between 14 and 16 years of age. 550 children remain in the study, which will continue until the last children have reached the age of 20 years.

ELIGIBILITY:
Inclusion Criteria:

* children at the age of 7 months and their families, recruited from the general population

Exclusion Criteria:

* severe sickness

Ages: 7 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1062
Dates: Start 1990-05; Study Completion 2005-08

PRIMARY OUTCOMES:
Intake of nutrients
Serum lipid and lipoprotein concentrations
Growth and development
Smoking
Physical activity level and fitness
Intima-media thickness of arteries and rate of NO-induced vasodilatation

SECONDARY OUTCOMES:
Psychological burden caused by the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Olli G Simell, MD, PhD, Principal Investigator — University of Turku, Turku, Finland
Locations (1):
- Department of Pediatrics, University of Turku, Turku, Finland

REFERENCES:
- [Background] Angle S, Keskinen S, Lapinleimu H, Helenius H, Raittinen P, Ronnemaa T, Simell O. Weight gain since infancy and prepubertal body dissatisfaction. Arch Pediatr Adolesc Med. 2005 Jun;159(6):567-71. doi: 10.1001/archpedi.159.6.567. PMID 15939857
- [Background] Viikari JS, Niinikoski H, Juonala M, Raitakari OT, Lagstrom H, Kaitosaari T, Ronnemaa T, Simell O. Risk factors for coronary heart disease in children and young adults. Acta Paediatr Suppl. 2004 Dec;93(446):34-42. doi: 10.1111/j.1651-2227.2004.tb00237.x. PMID 15702668
- [Background] Volanen I, Raitakari OT, Vainionpaa R, Arffman M, Aarnisalo J, Angle S, Kallio K, Simell O. Serum lipid profiles poorly correlate with Chlamydia pneumoniae, Helicobacter pylori, and cytomegalovirus seropositivity in prospectively followed-up healthy children. Arterioscler Thromb Vasc Biol. 2005 Apr;25(4):827-32. doi: 10.1161/01.ATV.0000158382.50942.6a. Epub 2005 Feb 3. PMID 15692096
- [Background] Hakanen M, Ronnemaa T, Talvia S, Rask-Nissila L, Koulu M, Viikari J, Bergendahl M, Simell O. Serum leptin concentration poorly reflects growth and energy and nutrient intake in young children. Pediatrics. 2004 May;113(5):1273-8. doi: 10.1542/peds.113.5.1273. PMID 15121941
- [Background] Ruottinen S, Karjalainen S, Pienihakkinen K, Lagstrom H, Niinikoski H, Salminen M, Ronnemaa T, Simell O. Sucrose intake since infancy and dental health in 10-year-old children. Caries Res. 2004 Mar-Apr;38(2):142-8. doi: 10.1159/000075938. PMID 14767171
- [Derived] Heiskanen MA, Aatsinki A, Hakonen P, Kartiosuo N, Munukka E, Lahti L, Keskitalo A, Huovinen P, Niinikoski H, Viikari J, Ronnemaa T, Lagstrom H, Jula A, Raitakari O, Rovio SP, Pahkala K. Association of Long-Term Habitual Dietary Fiber Intake since Infancy with Gut Microbiota Composition in Young Adulthood. J Nutr. 2024 Feb;154(2):744-754. doi: 10.1016/j.tjnut.2024.01.008. Epub 2024 Jan 12. PMID 38219864
- [Derived] Laitinen TT, Saha E, Pahkala K, Kartiosuo N, Nuotio J, Lagstrom H, Viikari J, Ronnemaa T, Jula A, Raitakari O, Niinikoski H. Associations of breastfeeding duration with serum lipid values from infancy until age 20 years - the STRIP study. Scand J Public Health. 2024 Aug;52(6):685-691. doi: 10.1177/14034948231183030. Epub 2023 Jun 30. PMID 37387272
- [Derived] Laitinen TT, Nuotio J, Niinikoski H, Juonala M, Rovio SP, Viikari JSA, Ronnemaa T, Magnussen CG, Sabin M, Burgner D, Jokinen E, Lagstrom H, Jula A, Simell O, Raitakari OT, Pahkala K. Attainment of Targets of the 20-Year Infancy-Onset Dietary Intervention and Blood Pressure Across Childhood and Young Adulthood: The Special Turku Coronary Risk Factor Intervention Project (STRIP). Hypertension. 2020 Nov;76(5):1572-1579. doi: 10.1161/HYPERTENSIONAHA.120.15075. Epub 2020 Sep 14. PMID 32921196
- [Derived] Laitinen TT, Nuotio J, Rovio SP, Niinikoski H, Juonala M, Magnussen CG, Jokinen E, Lagstrom H, Jula A, Viikari JSA, Ronnemaa T, Simell O, Raitakari OT, Pahkala K. Dietary Fats and Atherosclerosis From Childhood to Adulthood. Pediatrics. 2020 Apr;145(4):e20192786. doi: 10.1542/peds.2019-2786. Epub 2020 Mar 24. PMID 32209700
- [Derived] Laitinen TT, Nuotio J, Juonala M, Niinikoski H, Rovio S, Viikari JSA, Ronnemaa T, Magnussen CG, Jokinen E, Lagstrom H, Jula A, Simell O, Raitakari OT, Pahkala K. Success in Achieving the Targets of the 20-Year Infancy-Onset Dietary Intervention: Association With Insulin Sensitivity and Serum Lipids. Diabetes Care. 2018 Oct;41(10):2236-2244. doi: 10.2337/dc18-0869. Epub 2018 Aug 2. PMID 30072407
- [Derived] Lehtovirta M, Pahkala K, Niinikoski H, Kangas AJ, Soininen P, Lagstrom H, Viikari JSA, Ronnemaa T, Jula A, Ala-Korpela M, Wurtz P, Raitakari OT. Effect of Dietary Counseling on a Comprehensive Metabolic Profile from Childhood to Adulthood. J Pediatr. 2018 Apr;195:190-198.e3. doi: 10.1016/j.jpeds.2017.11.057. Epub 2018 Feb 1. PMID 29397160
- [Derived] Jaakkola JM, Pahkala K, Ronnemaa T, Viikari J, Niinikoski H, Jokinen E, Lagstrom H, Jula A, Raitakari O. Longitudinal child-oriented dietary intervention: Association with parental diet and cardio-metabolic risk factors. The Special Turku Coronary Risk Factor Intervention Project. Eur J Prev Cardiol. 2017 Nov;24(16):1779-1787. doi: 10.1177/2047487317720286. Epub 2017 Jul 20. PMID 28727955
- [Derived] Mikola H, Pahkala K, Niinikoski H, Ronnemaa T, Viikari JSA, Jula A, Juonala M, Raitakari OT. Cardiometabolic Determinants of Carotid and Aortic Distensibility From Childhood to Early Adulthood. Hypertension. 2017 Aug;70(2):452-460. doi: 10.1161/HYPERTENSIONAHA.117.09027. Epub 2017 Jun 26. PMID 28652463
- [Derived] Jaasaari P, Tolvanen M, Niinikoski H, Karjalainen S. Advanced dental maturity of Finnish 6- to 12-yr-old children is associated with high energy intake. Eur J Oral Sci. 2016 Oct;124(5):465-471. doi: 10.1111/eos.12292. Epub 2016 Sep 20. PMID 27644174
- [Derived] Jaakkola JM, Pahkala K, Viitala M, Ronnemaa T, Viikari J, Niinikoski H, Lagstrom H, Jula A, Simell O, Raitakari O. Association of Adiponectin with Adolescent Cardiovascular Health in a Dietary Intervention Study. J Pediatr. 2015 Aug;167(2):353-60.e1. doi: 10.1016/j.jpeds.2015.04.044. Epub 2015 May 15. PMID 25982143
- [Derived] Lapinleimu J, Raitakari OT, Lapinleimu H, Pahkala K, Ronnemaa T, Simell OG, Viikari JS. High lipoprotein(a) concentrations are associated with impaired endothelial function in children. J Pediatr. 2015 Apr;166(4):947-52.e1-2. doi: 10.1016/j.jpeds.2014.12.051. Epub 2015 Feb 4. PMID 25661407
- [Derived] Nupponen M, Pahkala K, Juonala M, Magnussen CG, Niinikoski H, Ronnemaa T, Viikari JS, Saarinen M, Lagstrom H, Jula A, Simell O, Raitakari OT. Metabolic syndrome from adolescence to early adulthood: effect of infancy-onset dietary counseling of low saturated fat: the Special Turku Coronary Risk Factor Intervention Project (STRIP). Circulation. 2015 Feb 17;131(7):605-13. doi: 10.1161/CIRCULATIONAHA.114.010532. Epub 2015 Jan 20. PMID 25605660
- [Derived] Ahola-Olli AV, Pitkanen N, Kettunen J, Oikonen MK, Mikkila V, Lehtimaki T, Kahonen M, Pahkala K, Niinikoski H, Kangas AJ, Soininen P, Ala-Korpela M, Viikari JS, Ronnemaa T, Simell O, Raitakari OT. Interactions between genetic variants and dietary lipid composition: effects on circulating LDL cholesterol in children. Am J Clin Nutr. 2014 Dec;100(6):1569-77. doi: 10.3945/ajcn.114.085027. Epub 2014 Oct 8. PMID 25411292
- [Derived] Mikola H, Pahkala K, Ronnemaa T, Viikari JS, Niinikoski H, Jokinen E, Salo P, Simell O, Juonala M, Raitakari OT. Distensibility of the aorta and carotid artery and left ventricular mass from childhood to early adulthood. Hypertension. 2015 Jan;65(1):146-52. doi: 10.1161/HYPERTENSIONAHA.114.03316. Epub 2014 Oct 27. PMID 25350980
- [Derived] Laine MA, Tolvanen M, Pienihakkinen K, Soderling E, Niinikoski H, Simell O, Karjalainen S. The effect of dietary intervention on paraffin-stimulated saliva and dental health of children participating in a randomized controlled trial. Arch Oral Biol. 2014 Feb;59(2):217-25. doi: 10.1016/j.archoralbio.2013.11.013. Epub 2013 Dec 1. PMID 24370194
- [Derived] Oranta O, Pahkala K, Ruottinen S, Niinikoski H, Lagstrom H, Viikari JS, Jula A, Loo BM, Simell O, Ronnemaa T, Raitakari OT. Infancy-onset dietary counseling of low-saturated-fat diet improves insulin sensitivity in healthy adolescents 15-20 years of age: the Special Turku Coronary Risk Factor Intervention Project (STRIP) study. Diabetes Care. 2013 Oct;36(10):2952-9. doi: 10.2337/dc13-0361. Epub 2013 Jun 25. PMID 23801725
- [Derived] Pahkala K, Laitinen TT, Heinonen OJ, Viikari JS, Ronnemaa T, Niinikoski H, Helajarvi H, Juonala M, Simell O, Raitakari OT. Association of fitness with vascular intima-media thickness and elasticity in adolescence. Pediatrics. 2013 Jul;132(1):e77-84. doi: 10.1542/peds.2013-0041. Epub 2013 Jun 10. PMID 23753102
- [Derived] Pahkala K, Hietalampi H, Laitinen TT, Viikari JS, Ronnemaa T, Niinikoski H, Lagstrom H, Talvia S, Jula A, Heinonen OJ, Juonala M, Simell O, Raitakari OT. Ideal cardiovascular health in adolescence: effect of lifestyle intervention and association with vascular intima-media thickness and elasticity (the Special Turku Coronary Risk Factor Intervention Project for Children [STRIP] study). Circulation. 2013 May 28;127(21):2088-96. doi: 10.1161/CIRCULATIONAHA.112.000761. Epub 2013 Apr 23. PMID 23613255
- [Derived] Niinikoski H, Ruottinen S. Is carbohydrate intake in the first years of life related to future risk of NCDs? Nutr Metab Cardiovasc Dis. 2012 Oct;22(10):770-4. doi: 10.1016/j.numecd.2012.05.002. Epub 2012 Jul 11. PMID 22789807
- [Derived] Niinikoski H, Pahkala K, Ala-Korpela M, Viikari J, Ronnemaa T, Lagstrom H, Jokinen E, Jula A, Savolainen MJ, Simell O, Raitakari OT. Effect of repeated dietary counseling on serum lipoproteins from infancy to adulthood. Pediatrics. 2012 Mar;129(3):e704-13. doi: 10.1542/peds.2011-1503. Epub 2012 Feb 13. PMID 22331346
- [Derived] Pahkala K, Heinonen OJ, Simell O, Viikari JS, Ronnemaa T, Niinikoski H, Raitakari OT. Association of physical activity with vascular endothelial function and intima-media thickness. Circulation. 2011 Nov 1;124(18):1956-63. doi: 10.1161/CIRCULATIONAHA.111.043851. Epub 2011 Oct 3. PMID 21969011
- [Derived] Karjalainen S, Soderling E, Saarinen M, Larsson B, Johansson I, Simell O, Niinikoski H. Effect of infancy-onset dietary intervention on salivary cholesterol of children: a randomized controlled trial. J Dent Res. 2011 Jul;90(7):868-73. doi: 10.1177/0022034511405328. Epub 2011 Apr 7. PMID 21474838
- [Derived] Kallio K, Jokinen E, Saarinen M, Hamalainen M, Volanen I, Kaitosaari T, Ronnemaa T, Viikari J, Raitakari OT, Simell O. Arterial intima-media thickness, endothelial function, and apolipoproteins in adolescents frequently exposed to tobacco smoke. Circ Cardiovasc Qual Outcomes. 2010 Mar;3(2):196-203. doi: 10.1161/CIRCOUTCOMES.109.857771. Epub 2010 Mar 2. PMID 20197510
- [Derived] Niinikoski H, Jula A, Viikari J, Ronnemaa T, Heino P, Lagstrom H, Jokinen E, Simell O. Blood pressure is lower in children and adolescents with a low-saturated-fat diet since infancy: the special turku coronary risk factor intervention project. Hypertension. 2009 Jun;53(6):918-24. doi: 10.1161/HYPERTENSIONAHA.109.130146. Epub 2009 Apr 13. PMID 19364991
- [Derived] Hakanen M, Raitakari OT, Lehtimaki T, Peltonen N, Pahkala K, Sillanmaki L, Lagstrom H, Viikari J, Simell O, Ronnemaa T. FTO genotype is associated with body mass index after the age of seven years but not with energy intake or leisure-time physical activity. J Clin Endocrinol Metab. 2009 Apr;94(4):1281-7. doi: 10.1210/jc.2008-1199. Epub 2009 Jan 21. PMID 19158205
- [Derived] Volanen I, Kallio K, Saarinen M, Jarvisalo MJ, Vainionpaa R, Ronnemaa T, Viikari J, Marniemi J, Simell O, Raitakari OT. Arterial intima-media thickness in 13-year-old adolescents and previous antichlamydial antimicrobial use: a retrospective follow-up study. Pediatrics. 2008 Sep;122(3):e675-81. doi: 10.1542/peds.2008-0220. PMID 18762502
- [Derived] Ruottinen S, Niinikoski H, Lagstrom H, Ronnemaa T, Hakanen M, Viikari J, Jokinen E, Simell O. High sucrose intake is associated with poor quality of diet and growth between 13 months and 9 years of age: the special Turku Coronary Risk Factor Intervention Project. Pediatrics. 2008 Jun;121(6):e1676-85. doi: 10.1542/peds.2007-1642. PMID 18519471
- [Derived] Kallio K, Jokinen E, Raitakari OT, Hamalainen M, Siltala M, Volanen I, Kaitosaari T, Viikari J, Ronnemaa T, Simell O. Tobacco smoke exposure is associated with attenuated endothelial function in 11-year-old healthy children. Circulation. 2007 Jun 26;115(25):3205-12. doi: 10.1161/CIRCULATIONAHA.106.674804. Epub 2007 Jun 4. PMID 17548727